CLINICAL TRIAL: NCT05104177
Title: Effectivness of Conservative Techniques in Management of PAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Heshmat Atrees Mohammed, Principal investigator, Assiut University
Other Study IDs: conservative techniques in PAS
Record Dates: First submitted 2021-10-09; First posted 2021-11-02 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: conservative tecchniques in management of PAS — Meticulous complete dissection of the urinary bladder from the lower uterine segment.
  * Transverse uterine incision above the visible vascular bulge if visible in cases with anterior PAS, otherwise a transverse lower uterine segment incision is performed in the same site of previous CS scar.
  * Delivery of the baby, clamping of the cord and administration IV 10 IU oxytocin.
  * Bilateral uterine artery ligation at one or two levels below the lowermost part of the placenta.
  * Removal of the separable part of the placenta from above downwards, until the adherent part is encountered.
  * A decision is taken to either resect a wedge of the myometrium above the adherent placenta (in case the adherent area is small and anterior), or removing all the adherent placenta then inserting a rubber or plastic catheter inside the cervical canal then identifying and closing the placental pouch. Care is given to rapidly perform this step to decrease the blood loss after removing the placenta

SUMMARY:
To evaluate the effectiveness of conservative techniques for placenta accreta spectrum to reduce maternal mortality and morbidity

DETAILED DESCRIPTION:
Placenta accreta spectrum (PAS) represents the spectrum of clinical conditions when part or whole of the placenta becomes abnormally adherent or invades the myometrium . Over the last 40 years, caesarean delivery rates around the world have risen from less than 10% to over 30%, and almost simultaneously a 10-fold increase in the incidence of PAS . PAS is one of the most dangerous conditions of the pregnancy as it is significantly associated with maternal morbidity and mortality .

Ultrasound imaging is the most commonly used technique to diagnose PAS disorders prenatally. There is also wide variation globally on the management of PAS disorders, with some centres opting for a radical approach, whereas others have proposed a range of conservative approaches .

The conservative approaches include one-step conservative surgery, leaving the placenta in situ, the Triple-P procedure, and transverse B-Lynch suture . Recently, Women's health hospital has adopted a new approach for conservative management of most cases of PAS, including wedge resection of the myometrium over the adherent part of the placenta, or a staged-approach following delivery of the fetus starting with meticulous dissection of the urinary bladder form the lower uterine segment, then bilateral uterine artery ligation at a level below the apparent placenta-myometrial bulge, followed by removal of the placenta, after which a catheter is inserted in the cervix and the placental pouch is closed .

ELIGIBILITY:
Inclusion Criteria:

1. - Gestational age starting from 28 weeks onwards.
2. - Women with at least 1 previous hysterotomy (e.g. Caesarean deliveries, myomectomy)
3. - Elective or emergent Caesarean deliveries

Exclusion Criteria:

* A pre-existing decision of performing intrapartum hysterectomy

Ages: 19 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — females in reproductive age
Study Population: females in reproductive age
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
number of patients who undergo hysterectomy after failure of conservative techniques | baseline
  Counting patients who undergo hystrectomy after conservative techniques to evalute it's effectivness

SECONDARY OUTCOMES:
recurrence of PAS | baseine
  Nomber of cases recurrence who will have of PAS In subsequent pregnancies after conservative techniques

REFERENCES:
- [Background] Jauniaux E, Collins S, Burton GJ. Placenta accreta spectrum: pathophysiology and evidence-based anatomy for prenatal ultrasound imaging. Am J Obstet Gynecol. 2018 Jan;218(1):75-87. doi: 10.1016/j.ajog.2017.05.067. Epub 2017 Jun 24. PMID 28599899